CLINICAL TRIAL: NCT02219412
Title: An Open Label, Two Arms, Randomized Controlled Pilot Study Comparing the Arachidonic Acid-induced Platelet Aggregation Rate in Patients With Stable Coronary Artery Disease Treated With Ticagrelor Monotherapy or Ticagrelor and Asprin
Brief Title: Arachidonic Acid-induced Platelet Aggregation Rate in Patients With Stable CAD Treated With Ticagrelor Monotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yong Huo (Other)
Responsible Party: Sponsor-Investigator, Yong Huo, The director of the Department of Cardiology and heart center of Peking University First Hospital, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSBRIL0235
Record Dates: First submitted 2014-07-24; First posted 2014-08-18 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Coronary Heart Disease
Keywords: ticagrelor; platelet aggregation rate; ADP antagonist; antiplatelet therapy
MeSH Terms: conditions — Coronary Disease | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ticagrelor mono-therapy (Experimental): Take ticagrelor 90 mg Bid for 2 weeks.
  Interventions: Drug: ticagrelor
- aspirin/ticagrelor dual-therapy (Active Comparator): Take ticagrelor 90mg Bid plus Aspirin 100mg Qd and treated for 2 weeks.
  Interventions: Drug: ticagrelor; Drug: Aspirin

INTERVENTIONS:
Drug: ticagrelor — 90 mg bid for 2 weeks
  Other Names: Brilinta
Drug: Aspirin — 100mg Qd for 2 weeks.
  Arms: aspirin/ticagrelor dual-therapy

SUMMARY:
This study was a feasibility trial that was designed to provide preliminary observations and generate hypotheses for future studies. The aim of the study is to estimate the difference of arachidonic acid induced platelet aggregation rate between ticagrelor mono-therapy and aspirin/ticagrelor dual-therapy after 14 days of treatment in patients with stable coronary artery disease. The potential hypothesis is that the arachidonic acid (AA) induced platelet aggregation rate after 2 weeks of ticagrelor mono-therapy is comparable to that of aspirin/ticagrelor dual-therapy.

DETAILED DESCRIPTION:
This is a randomized, open labeled, active-controlled pilot study to estimate the difference of arachidonic acid induced platelet aggregation rate between ticagrelor monotherapy and aspirin/ticagrelor dual-therapy in patients with stable coronary heart disease. The anticipated duration of the study is approximately 9 months, including an anticipated enrolment period of 8 months and follow-up period of 4weeks.

Patients with documented coronary heart disease and currently receiving dual-antiplatelet therapy with standard dose aspirin and clopidogrel will be enrolled from the study site. For patients post acute coronary syndrome (ACS) or percutaneous coronary intervention (PCI), they must be on dual-antiplatelet therapy for at least 12 months to be eligible for the study.

The study plan, including enrolment/randomization and follow-up visits, is outlined in Table 1. Eligible patients will enter a washout phase with ticagrelor for 2 weeks. Then they will be randomized to take either ticagrelor alone or aspirin/ticagrelor for 14 days. The efficacy evaluation will be done at 7 and 14days after randomization. The primary efficacy parameter is the rate of arachidonic acid induced platelet aggregation after 14 days of treatment. All patients will be treated to standards of care for coronary heart disease secondary prevention.

Visit 0 (Screening and Enrollment, 0 day) All potentially eligible patients will undergo a screening visit following their signed informed consent.

Following an 8-hour fast, the patients will have screening evaluations performed. Demography, medical history, and concomitant medication will be recorded. A physical examination and vital signs(pulse and BP), height and weight, as well as blood sampling for laboratory assessments of complete blood count (CBC) with differential, serum creatinine, alanine aminotransferase (ALT) and aspartate aminotransferase (AST), and AA, adenosine diphosphate (ADP) and collagen induced platelet aggregation rate will be done. Standard 12-lead electrocardiogram (ECG) readings will be recorded.

Patients meeting all inclusion criteria and with no exclusion criteria will be enrolled. Patients will receive ticagrelor mono-therapy from the evening for 14 days. IP will be dispensed.

Visit 1 (Randomization, 14 days) Suspected adverse events (AEs) will be recorded. A physical examination and vital signs (pulse and BP), as well as blood sampling for laboratory assessments of AA, ADP and collagen induced platelet aggregation rate and serum thromboxane B2 concentration will be done.

Patients should be told to take ticagrelor in the morning of Visit 1. Patients will be randomized in a 1:1 ratio to receive either ticagrelor mono-therapy or aspirin/ticagrelor dual-therapy. Investigational product (IP) will be returned and compliance assessed and new bottles of IP will be dispensed according to randomized groups.

Visit 2 (21 days) Suspected AEs will be recorded. Vital signs (pulse and BP) as well as blood sampling for laboratory assessments of AA, ADP and collagen induced platelet aggregation rate will be done.

Visit 3 (End of treatment, 28 days) Suspected AEs will be recorded. Vital signs (pulse and BP) as well as blood sampling for laboratory assessments of CBC with differential, Scr, ALT and AST, AA, ADP and collagen induced platelet aggregation rate will be done. IP will be returned and compliance assessed. Instructions for medication after study will be given to patients at this time.

For patients who prematurely discontinued the randomized treatment, a complete end of treatment visit will be preferred.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Aged >18 years.
* Documented stable coronary artery disease.
* Currently receiving dual-antiplatelet therapy with aspirin 100mg/d and clopidogrel 75mg/d.

Exclusion Criteria:

* History of acute coronary syndrome within 12 months of screening.
* History of percutaneous coronary intervention within 12 months of screening.
* Any indication (eg, atrial fibrillation,prosthetic heart valve, or coronary stent) for antithrombotic therapy(eg, warfarin, clopidogrel, or aspirin dose other than 75 to 100 mg/during the study period).
* AA induced platelet aggregation rate >20% on aspirin+clopidogrel measured by light transmission platelet aggregation test with the past 3 months.
* Congestive heart failure or left ventricular ejection fraction <35%.
* Forced expiratory volume in the first second forced vital capacity below the lower limits of normal.
* Bleeding diathesis or severe pulmonary disease.
* Active pathological bleeding.
* History of intracranial hemorrhage.
* Hypersensitivity to ticagrelor or any of the excipients.
* Severe hepatic impairment.
* Pregnancy.
* Current smoking.
* Platelet count <100 000/mm3 or hemoglobin <10 g/dL.
* HemoglobinA1c >10%.
* History of drug addiction or alcohol abuse in the past 2 years.
* Need for nonsteroidal anti-inflammatory drug.
* Creatinine clearance<30 mL/min.
* Concomitant therapy with moderate or strong cytochrome P450 3A inhibitors, substrates, or strong cytochrome P450 3A inducers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The rate of AA induced platelet aggregation | Day 14 after randomization
  The rate of AA induced platelet aggregation will be measured at day 14 after randomization.

SECONDARY OUTCOMES:
The rate of ADP induced platelet aggregation | Day 7 and day 14 after randomization
  The rate of ADP induced platelet aggregation will be measured at day 7 and day 14 after randomization.
The rate of collagen induced platelet aggregation | Day 7 and day 14 after randomization
  The rate of d collagen induced platelet aggregation will be measured at day 7 and day 14 after randomization.
The serum concentration of Thromboxane B2 | Day 7 and day 14 after randomization
  The serum concentration of Thromboxane B2 will be measured at day7 and day 14 after randomization
The rate of AA induced platelet aggregation | Day 7 after randomization
  The rate of collagen induced platelet aggregation will be measured on Day 7 after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Huo Yong, MD, Study Chair — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No